CLINICAL TRIAL: NCT05577338
Title: Neural Mechanism Underlying the Beneficial Effect of Theory of Mind Psychotherapy on Early-onset Schizophrenia: A Randomized Controlled Trial.
Brief Title: ToM Psychotherapy and Brain Networks in EOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PJ2022-10-37
Record Dates: First submitted 2022-09-19; First posted 2022-10-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2021-08

CONDITIONS: Early-onset Schizophrenia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- training group (Experimental): Theory of Mind psychotherapy psychotherapy
  Interventions: Behavioral: Theory of Mind psychotherapy
- active control group (Active Comparator): receive disease-related health knowledge
  Interventions: Behavioral: health education

INTERVENTIONS:
Behavioral: Theory of Mind psychotherapy — a semi-structured, multidomain, tailored group psychotherapy
  Arms: training group
Behavioral: health education — disease-related health knowledge
  Arms: active control group

SUMMARY:
Background: Presence of a series of typical physical symptoms is an enduring and functionally relevant feature of early-onset schizophrenia (EOS). Psychotherapy improves clinical symptoms in adults with schizophrenia, although data in adolescents with EOS remain scarce. The purpose of this study is to examine the efficacy of the adapted group psychotherapy in improving clinical symptoms from a perspective of neuroimaging in a sample of symptomatically stable adolescents with EOS.

Methods: Investigators conducted a double-blind randomized controlled trial using multidomain, adaptive, group psychotherapy in 28 EOS patients, who were randomly allocated into either training (group psychotherapy) or active control (health education) groups. Data of diffusion tensor imaging, and clinical symptoms were obtained at baseline and after an average of 2 hours/day, 2 days/week for 4 weeks of intervention.

DETAILED DESCRIPTION:
Schizophrenia is a chronic psychiatric disorder with a heterogeneous genetic and neurobiological background that influences early brain development and is expressed as a combination of psychotic symptoms - such as hallucinations, delusions and disorganization - and motivational and cognitive dysfunctions. Schizophrenia occurs worldwide, and for decades it was generally believed to have a uniform lifetime morbid risk of 1% across time, geography, and gender. Characteristic, a substantial proportion of patients with schizophrenia experience the onset of their illness by age 18, defined as early-onset schizophrenia (EOS) and were found to be associated with higher rates of premorbid abnormalities, worse cognitive performance and worse functional outcome compared to individuals with adult-onset schizophrenia. Recently, EOS patients have been the focus of substantial interest, since studies of patients with adolescent onset could provide insights into the development of the disorder, in particular the interaction between normal maturational processes and the disorder. Furthermore, EOS is featured as a debilitating form of schizophrenia that has poor prognosis and functional outcomes and that places heavy demands on caregivers.

To the best of investigators' knowledge that enduring cognitive impairment is a core feature of the illness that predict chronicity and contribute to poor functional outcomes. As EOS is potentially a key stage at which early intervention may delay or prevent the poor outcomes, and pharmacological interventions have a limited effect on cognitive impairment in EOS patients, there is a critical need and growing interest in psychosocial interventions for effective treatments for cognitive impairment in young persons with this condition, which are now recognized as an important component of a comprehensive therapeutic approach in schizophrenia. Recent advances in cognitive training, however, may inform strategies to treat EOS. For instance, as cognitive remediation therapy (CRT) uses scientific principles of learning to target cognitive deficits with the ultimate goal of improving functional outcome, there is now a substantial body of evidence in support of its efficacy in adults with schizophrenia. Furthermore, the adult recommendations are adopted in clinical practice for the treatment (referring to group psychotherapy in this study) of children and adolescents with psychosis, as there is a paucity of studies conducted exclusively with EOS patients.

The notion that specific cognitive and social abilities arise from functionally distinct brain regions has been proved by means of multimodal neuroimaging techniques mainly including structural and functional Magnetic Resonance Imaging (MRI). Previous studies of EOS patients have found abnormalities in white matter microstructure, slower white matter growth rates and disrupted functional connectivity in brain networks involved in sensorimotor processing, social cognitions and executive functions. The abovementioned evidence supports the neurodevelopmental and dis-connectivity hypotheses of schizophrenia, but the specific pattern of abnormal brain structural connectivity in EOS remains scarce. Graph-theory analysis, which examines the important properties of complex systems (i.e., centrality, global efficiency, local efficiency and small-world property), is a useful tool to quantify the topology of abnormal brain networks in EOS. To our knowledge, using the graph-based network approach, previous research has mapped structural networks in adult patients with schizophrenia based on across-subject covariance in morphological indexes, such as cortical thickness, gyrification and grey matter volumes. However, in this context, investigators constructed structural connections of brain networks characterized by white matter integrity measured by diffusion tensor imaging (DTI). Moreover, it remains unclear that how brain structural topology is altered in EOS patients after the intervention of group psychotherapy.

In this study, investigators conducted an adaptable randomized controlled trial (RCT) to investigate the effects of group psychotherapy on brain structural connectivity in EOS patients using a graph-based approach of DTI. Investigators hypothesized that adaptable group psychotherapy would help to preserve brain structural network connectivity in addition to better ameliorating clinical symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of EOS
* Right-handed subjects
* Aged 13 - 18 years old
* Capable of understanding, judgments and expression

Exclusion Criteria:

* The presence of other psychiatric disorders such as substance-induced mood disorder, bipolar disorders, anxiety disorders, substance abuse, or dependence
* A history of significant physical or neurological disease
* A history of head injury with loss of consciousness
* A history of electroconvulsive therapy
* Contraindications for MRI such as claustrophobia
* Mental retardation.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
changes in positive and negative scale score (PANSS) | Change from Baseline PANSS at 1 month
  A standardized rating scale of clinical questionnaires without units designed to assess the severity of symptoms of different types of schizophrenia.
changes in binary betweenness centrality | Change from Baseline binary betweenness centrality at 1 month
  One of the brain structural network properties computed via the software packages Brain functional Magnetic Resonance Imaging (FMRIB) Software Library (FSL3) and Diffusion Toolkit (DTK4) without units and captures the extent to which a node is in-between several other nodes in a network.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

REFERENCES:
- [Background] Kumra S, Charles Schulz S. Editorial: research progress in early-onset schizophrenia. Schizophr Bull. 2008 Jan;34(1):15-7. doi: 10.1093/schbul/sbm123. Epub 2007 Nov 28. PMID 18048380
- [Background] Vernal DL, Boldsen SK, Lauritsen MB, Correll CU, Nielsen RE. Long-term outcome of early-onset compared to adult-onset schizophrenia: A nationwide Danish register study. Schizophr Res. 2020 Jun;220:123-129. doi: 10.1016/j.schres.2020.03.045. Epub 2020 Apr 13. PMID 32299717
- [Background] Armando M, Pontillo M, Vicari S. Psychosocial interventions for very early and early-onset schizophrenia: a review of treatment efficacy. Curr Opin Psychiatry. 2015 Jul;28(4):312-23. doi: 10.1097/YCO.0000000000000165. PMID 26001923
- [Background] Puig O, Penades R, Baeza I, De la Serna E, Sanchez-Gistau V, Bernardo M, Castro-Fornieles J. Cognitive remediation therapy in adolescents with early-onset schizophrenia: a randomized controlled trial. J Am Acad Child Adolesc Psychiatry. 2014 Aug;53(8):859-68. doi: 10.1016/j.jaac.2014.05.012. Epub 2014 Jun 21. PMID 25062593
- [Derived] Liu S, Zhong H, Qian Y, Cai H, Jia YB, Zhu J. Neural mechanism underlying the beneficial effect of Theory of Mind psychotherapy on early-onset schizophrenia: a randomized controlled trial. J Psychiatry Neurosci. 2023 Nov 7;48(6):E421-E430. doi: 10.1503/jpn.230049. Print 2023 Nov-Dec. PMID 37935475